CLINICAL TRIAL: NCT06269588
Title: A Prospective, Multi-center, Single-arm, Pilot Clinical Trial to Evaluate Efficacy and Safety of Nexpowder™ for Hemostatic Treatment of Non-variceal, Upper Gastrointestinal Bleeding
Brief Title: Efficacy and Safety of Nexpowder™ for Non-variceal, Upper Gastrointestinal Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Collaborators: Next Biomedical Co., Ltd. (Industry); Tan Tock Seng Hospital (Other); National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBM-NP004
Record Dates: First submitted 2023-10-19; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-10

CONDITIONS: Gastrointestinal Hemorrhage; Hematemesis; With Ulcer; Endoscopy
Keywords: gastrointestinal bleeding; hemostatic powder
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hematemesis

STUDY DESIGN:
Intervention Model Description: prospective single arm intervention cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic hemostasis using Nexpowder (Experimental): Subjects with non variceal upper GI bleeding will undergo nndoscopic hemostasis using Nexpowder as primary treatment
  Interventions: Device: Nexpowder

INTERVENTIONS:
Device: Nexpowder — Endoscopic hemostasis

SUMMARY:
The purpose of this pilot clinical trial is to confirm the efficacy and safety of Nexpowder™ for hemostasis in pilot cohort of patients with NVUGIB in Singapore

DETAILED DESCRIPTION:
24 subjects with non variceal bleeding will be enrolled. The efficacy and safety of Nexpowder™ as primary technique of endoscopci hemostasis will be assessed in this pi,ot study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged over 21 to 75 years
2. Patients with confirmed nonvariceal, upper gastrointestinal bleeding
3. Patients who voluntarily agree to the clinical trial with informed consent
4. Patients who willing and able to comply with the study protocol

Exclusion Criteria:

1. Patients with an uncorrected coagulation disorder (PLT<50*109/L, INR>2)
2. Patients who are known to be pregnant or in lactation
3. Patients who have received another endoscopic treatment for the same part of the body within the days preceding the study
4. Patients for whom endoscopic treatment is prohibited due to comorbidity
5. Patients for whom the 30-day follow-up period is impossible
6. Patients who have participated within the past month in other related clinical trials that could affect the results of the study
7. Other cases in which participation in the study is judged inappropriate by the investigators

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
endoscopic hemostasis | up to 24 hours
  endoscopic hemostasis success rate

SECONDARY OUTCOMES:
recurrent bleeding rate on second-look endoscopy | 24 hours
  recurrent bleeding rate on second-look endoscopy
hydrogel persistence rate at the bleeding site | 24 hours
  hydrogel persistence rate at the bleeding site
Recurrent bleeding within 30 days after endoscopic therapy | 30 days
  Recurrent bleeding within 30 days after endoscopic therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No